CLINICAL TRIAL: NCT04089176
Title: Carbetocin Versus Oxytocin for Prevention of Postcesarean Hemorrhage in Pregnant Women With High Risk Postpartum Hemorrhage: a Randomized Controlled Trial
Brief Title: Carbetocin Versus Oxytocin for Prevention of Postcesarean Hemorrhage in Pregnancy With High Risk for PPH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T.Sopida
Record Dates: First submitted 2019-04-28; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Postpartum Hemorrhage; Cesarean Section; High Risk Pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- protocal A (Active Comparator): Carbetocin versus placebo
  Interventions: Drug: Carbetocin; Drug: oxytocin
- protocal B (Active Comparator): Oxytocin versus placebo
  Interventions: Drug: Carbetocin; Drug: oxytocin

INTERVENTIONS:
Drug: Carbetocin — carbetocin 100 mcg + RLS solution 10 ml injected directly into the vein over 2 min
Drug: oxytocin — oxytocin 20 IU diluted in 1000 ml of RLS solution administered intravenously at rate 120 ml/hr x 8 hr

SUMMARY:
Objective: study efficacy of carbtocin versus oxytocin for prevention postpartum hemorrhage in high risk pregnancy who undergo cesarean section

DETAILED DESCRIPTION:
Randomized controlled clinical trial. Defined patient in two group. Primary outcome is evaluate additional drug use Secondary outcome is evaluated estimated blood loss, hemoglobin level

ELIGIBILITY:
Inclusion Criteria:

* previous history of postpartum hemorrhage
* polyhydramnios
* fetal macrosomia
* previous cesarean section
* grand multiparity
* intramural myoma
* chorioamnionitis
* prolonged premature rupture of membrane
* augmentation of labour

Exclusion Criteria:

* pregnancy induce hypertension
* on anticoagulant
* placenta previa or placenta percreta

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Additional drug use | during intra-operation
  Number of additional drug use after intervention drug

SECONDARY OUTCOMES:
Estimate blood loss | During intra-opeartion and acute post operation period as 24 hours post operation
  amount of blood loss
Side effect | During intra-opeartion and acute post operation period as 24 hours post operation
  type of side effect
Hemoglobin level | Pre-operation and 24 hours post operation
  differentiation of hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand